CLINICAL TRIAL: NCT03714126
Title: A Non-Intervantional Study to Create a Patient Recordings and Clinical Database Using the Cordio System
Brief Title: Remote Speech Analysis in HF Patients Undergoing Haemodialysis
Status: Completed | Type: Observational
Sponsor: Cordio Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: CLN0014
Record Dates: First submitted 2018-10-17; First posted 2018-10-22 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2020-04

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HF patients: HF patients will use the Cordio Medical app to record in their hospital visits and at home.
  Interventions: Device: Cordio Medical

INTERVENTIONS:
Device: Cordio Medical — Recording to an app, no interference to the regular care

SUMMARY:
This is an observational, non-interventional, prospective, single-arm, open study for database establishment for R&D purposes. The study will be conducted in 1 site in Israel with up to fifty (50) patients. Patients under hemodialysis supervision will be enrolled in the clinical trial. Clinical information for the study will be collected at the hospital and at home. The patient will conduct recordings at home every day.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing hemodialysis every 5-10 days in order to balance their volume overload.
* Class C Heart Failure patient with reduced EF CHF (EF<40%) and NYHA 2-3.
* Patients with dyspnea clinically related to pulmonary congestion
* Patient with more than 3 months HF disease duration.
* The patient is willing to participate as evidenced by signing the written informed consent.
* Male or non-pregnant female patient

Exclusion Criteria:

* Subject who, in the Investigator's opinion, unable to comply with the daily use of the App due to mental disorders (e.g., depression, dementia).
* Patient who has had a major cardiovascular event (e.g., myocardial infraction, stroke) within 3 months prior to screening visit.
* Patients likely to undergo heart transplantation/ LVAD within 6 months of Screening Visit or baseline functional capacity of NYHA 4.
* Patients with evidence of active Infection.
* Patient with severe alcohol or drug use.
* Psychological instability, inappropriate attitude or motivation.
* Patient with life threatening debilitating disease other than cardiac.
* Subject currently enrolled in another investigational device or drug trial that has not completed the primary endpoint or that clinically interferes with the current study endpoints.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Acute and Chronic Congestive Heart Failure patients, undergoing hemodialysis in order to balance their volume overload.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2021-03-08 (Actual); Study Completion 2021-03-08 (Actual)

PRIMARY OUTCOMES:
Number of CHF patients with and without acute lung accumulation. in R&D Database | throughout study, upto 60 days per patient
  The objective of the study is to create a recordings database of CHF patients with and without acute lung accumulation.

CONTACTS AND LOCATIONS:
Overall Officials: Ittamar Gork, Dr., Principal Investigator — Hadassah Ein Kerem
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No